CLINICAL TRIAL: NCT01668277
Title: Effects of Hypertonic Saline on the Pulmonary Circulation in Children
Brief Title: Effects of Saline on Circulation in Children
Status: Terminated | Phase: Phase 2 | Type: Interventional
Sponsor: The Hospital for Sick Children (Other)
Responsible Party: Principal Investigator, Katherine Taylor, Staff Anesthesiologist, The Hospital for Sick Children
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 1000026525
Record Dates: First submitted 2012-08-08; First posted 2012-08-20 (Estimated); Last update posted 2020-11-02 (Actual); Status verified 2020-10

CONDITIONS: Pulmonary Hypertensive Crisis
Keywords: Pulmonary Hypertensive Crisis; Pediatrics; Hypertonic Saline
MeSH Terms: interventions — Saline Solution

STUDY DESIGN:
Who Masked: Investigator
Oversight: Data Monitoring Committee: No

ARMS (3):
- 3 ml/kg 7.2% NaCl (Experimental): The test fluids 7.2% NaCl 3 ml/kg will be infused over 10 min. The hemodynamic parameters will be determined before and after infusion by a cardiologist blinded to the type of infusion.
  Interventions: Drug: 7.2% NaCl
- 3 ml/kg 0.9% NaCl (Active Comparator): The test fluids 0.9% NaCl 3 ml/kg will be infused over 10 min. The hemodynamic parameters will be determined before and after infusion by a cardiologist blinded to the type of infusion.
  Interventions: Drug: 0.9% NaCl
- 20 ml/kg 0.9% NaCl (Active Comparator): The test fluids 0.9% NaCl 20 ml/kg will be infused over 10 min. The hemodynamic parameters will be determined before and after infusion by a cardiologist blinded to the type of infusion.
  Interventions: Drug: 0.9% NaCl

INTERVENTIONS:
Drug: 7.2% NaCl
  Arms: 3 ml/kg 7.2% NaCl
Drug: 0.9% NaCl
  Arms: 20 ml/kg 0.9% NaCl; 3 ml/kg 0.9% NaCl

SUMMARY:
Pulmonary hypertensive crisis is a life-threatening condition, in which the blood pressure in the pulmonary artery, vein, and capillaries. Infusion of hypertonic saline solutions expand the circulating volume, thus allowing more blood to flow and reducing pressure in the artery, vein, and capillaries. Furthermore, infusion of hypertonic saline has been shown to reduce both systemic and pulmonary vascular resistances in adults. If the pulmonary vascular resistance decreases more or to the same degree as the systemic resistance, infusion of hypertonic saline may prove beneficial in the treatment of pulmonary hypertensive crisis. The primary objective of this study is to investigate how a clinically relevant dose of hypertonic saline affects the systemic and pulmonary circulations in children undergoing cardiac catheterization during general anesthesia. This study hypothesizes that an infusion of hypertonic saline over 10 minutes will reduce the pulmonary vascular resistance more than the systemic vascular resistance.

ELIGIBILITY:
Inclusion Criteria:

* Children who have had a heart transplant and are scheduled for elective endomyocardial biopsies during general anaesthesia
* Age > 2 years

Exclusion Criteria:

* Plasma Na < 130 mmol/l or >150 mmol/l
* Refusal of consent
* An estimated pulmonary arterial pressure which is greater than or equal to 66% of systemic blood pressure
* Children with heart failure (right and/or left), i.e clinical suspicion by either a cardiologist or an anesthesiologist of inability to tolerate a fluid bolus of 3 ml/kg 7.2% NaCl corresponding to an expansion of the circulatory volume by approximately 9% (see the section on safety), which is the equivalent of infusion approximately 20 ml/kg 0.9% NaCl over 10 minutes.

Ages: 2 Years to 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 15 (Actual)
Dates: Start 2012-08; Primary Completion 2014-12 (Actual); Study Completion 2014-12 (Actual)

PRIMARY OUTCOMES:
Pulmonary Vascular Resistance Index | Change from Baseline in Pulmonary Vascular Resistance Index after 1 hour
  Pulmonary vascular resistance index, a hemodynamic measurement, will be performed during the cardiac catherization.
Systemic Vascular Resistance Index | Change from Baseline in Systemic Vascular Resistance Index after 1 hour
  Systemic vascular resistance index, a hemodynamic measurement, will be performed during the cardiac catherization.
Cardiac Index | Change from Baseline in Cardiac Index after 1 hour
  Cardiac index, a hemodynamic measurement, will be performed during the cardiac catherization.

SECONDARY OUTCOMES:
Blood Gas | Average over 1 hour
  Effect on blood hemoglobin, plasma potassium and sodium, measured on a blood gas analyzer
Plasma Volume | Average over 1 hour
  Effect on plasma volume calculated from the change in blood hemoglobin
Atrial Natriuretic Peptide | Average over 1 hour
  Effect on atrial natriuretic peptide

CONTACTS AND LOCATIONS:
Overall Officials: Katherine Taylor, MD, Principal Investigator — The Hospital for Sick Children
Locations (2):
- Canada (2):
  - Hospital For Sick Children, Toronto, Ontario
  - The Hospital for Sick Children, Toronto, Ontario